CLINICAL TRIAL: NCT04705493
Title: Validation of Uncalibrated Cardiac Output Measurement With LiDCOrapid in the Resuscitation of Critically Ill Patients With Septic Shock: A Prospective Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magdy Abdelmohsen Elsayed Mohamed, MSC, Cairo University
Other Study IDs: MD-84-2019
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Output, LIDCO Rapid, Septic Shock
Keywords: cardiac output , LIDCO . Septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Crystalloid Solutions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASE GROUP: Lidco rapid examination and echo examination were done to septic shock patients then the passive leg raising test was done and fluid responder cases were given mini fluid challenge and fluid challenge
  Interventions: Other: fluid resuscitation with crystalloid

INTERVENTIONS:
Other: fluid resuscitation with crystalloid — give two-volume of fluids initial 250ml then another 250 ml

SUMMARY:
Transthoracic echocardiography (TTE) has been used as a reference technique for CO measurement and its accuracy has been adequate for many clinical uses. TTE is painless, safe and non-invasive. Some drawbacks of TTE are being expensive, bulky and needs advanced training.

Currently, due to increased interest in minimally invasive hemodynamic monitoring, multiple new methods have become commercially available to assess CO: the arterial pulse aortic flow, bioreactance, and bioimpedance.

One of these new devices is LiDCOrapid (LiDCO Ltd, Cambridge, UK). It is a new, minimally invasive monitor which estimates beat-by-beat CO and fluid responsiveness from the arterial waveform.

It has been validated after vascular, urological and thoracic surgery and shows good agreement with the PA catheter in swine, in patients with normal left ventricular systolic function and in patients with vasodilatation. However, LiDCO has not yet been validated in patients with septic shock. Therefore, the aim of this study is to validate LiDCOrapid parameters in septic shock patients using TTE derived parameters as the non-invasive reference.

DETAILED DESCRIPTION:
Obtaining a patient's cardiac output (CO) could contribute to optimized, safe hemodynamic control. Accurate CO measurements can serve as a guide for resuscitation therapy, catecholamine use, differential diagnosis, and intervention during a circulatory failure. Although the thermodilution technique via a pulmonary artery catheter (PAC) has an invasive and intermittent, it remains the gold standard for CO measurements.

Previously monitoring of CO required invasive and costly devices limiting their use to intensive care setting. More recently ultrasound is increasingly being used and offers a range of non-invasive tools to estimate CO.

Transthoracic echocardiography (TTE) has been used as a reference technique for CO measurement and its accuracy has been adequate for many clinical uses. TTE is painless, safe and non-invasive. Some drawbacks of TTE are being expensive, bulky and needs advanced training.

Currently, due to increased interest in minimally invasive hemodynamic monitoring, multiple new methods have become commercially available to assess CO: the arterial pulse aortic flow, bioreactance, and bioimpedance.

One of these new devices is LiDCOrapid (LiDCO Ltd, Cambridge, UK). It is a new, minimally invasive monitor which estimates beat-by-beat CO and fluid responsiveness from the arterial waveform.

It has been validated after vascular, urological and thoracic surgery and shows good agreement with the PA catheter in swine, in patients with normal left ventricular systolic function and in patients with vasodilatation. However, LiDCO has not yet been validated in patients with septic shock. Therefore, the aim of this study is to validate LiDCOrapid parameters in septic shock patients using TTE derived parameters as the non-invasive reference.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Patients admitted to ICU with septic shock

Exclusion Criteria:

1. Patients with poor Echo window.
2. If they presented with a history of heart failure, valvular disease or arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed on any patient with septic shock admitted to the surgical ICU.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
primary outcome | on patient admission to the icu for 1 hour
  To measure cardiac output difference between LiDCOrapid measurement and echocardiographic measurement .

SECONDARY OUTCOMES:
secondary outcome | on patient admission to the icu for 1 hour
  to measure dose of vasopressors and inotropic agents
secondary outcome | on patient admission to the icu for 1 hour
  to measure heart rate
secondary outcome | on patient admission to the icu for 1 hour
  to measure stroke volume
secondary outcome | on patient admission to the icu for 1 hour
  to detect stroke volume variation
secondary outcome | on patient admission to the icu for 1 hour
  to record mean arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy Shcool of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided